CLINICAL TRIAL: NCT04921358
Title: A Randomized Phase 3 Study of Tislelizumab in Combination With Sitravatinib in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer That Progressed on or After Platinum-Based Chemotherapy and Anti-PD-(L)1 Antibody
Brief Title: Tislelizumab in Combination With Sitravatinib in Participants With Locally Advanced or Metastatic Non-Small Cell Lung Cancer
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Due to safety risks and unfavorable risk-benefit assessment results, the sponsor has decided to voluntarily terminate the study.
Sponsor: BeiGene (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BGB-A317-Sitravatinib-301; 2022-001779-15 (EudraCT Number); SAFFRON-301 (Other: BeiGene); CTR20211410/CTR20211409 (Other: ChinaDrugTrials)
Record Dates: First submitted 2021-05-25; First posted 2021-06-10 (Actual); Results first posted 2025-06-29 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Non-Small Cell Lung Cancer (NSCLC)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — tislelizumab; Docetaxel; sitravatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tislelizumab + Sitravatinib (Experimental): Participants received 200 mg of intravenous tislelizumab every 3 weeks, combined with 100 mg of oral sitravatinib daily until disease progression, intolerable toxicity, death, or withdrawal of consent, whichever occurred earlier.
  Interventions: Drug: Tislelizumab; Drug: Sitravatinib
- Docetaxel (Active Comparator): Participants received 75 mg/m² of intravenous docetaxel once every 3 weeks until disease progression, intolerable toxicity, death, or withdrawal of consent, whichever occurred earlier.
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Tislelizumab — 200 mg intravenously once every 3 weeks
  Other Names: BGB-A317
  Arms: Tislelizumab + Sitravatinib
Drug: Docetaxel — 75 mg/m^2 intravenously once every 3 weeks
  Arms: Docetaxel
Drug: Sitravatinib — 100 mg orally once daily
  Other Names: BGB-9468
  Arms: Tislelizumab + Sitravatinib

SUMMARY:
The purpose of this study was to evaluate the efficacy and safety of tislelizumab in combination with sitravatinib compared to docetaxel in participants with locally advanced or metastatic non-small cell lung cancer (NSCLC) who experienced disease progression following platinum-based chemotherapy and anti-programmed cell death protein-1 (PD-1)/programmed cell death ligand-1 (PD-L1) antibody treatment, with the anti-PD-(L)1 antibody administered either in combination with or sequentially before or after the platinum-based chemotherapy.

ELIGIBILITY:
Key Inclusion Criteria:

1. Metastatic or unresectable locally advanced histologically or cytologically confirmed Non-Small Cell Lung Cancer (NCSLC), not amenable to treatment with curative intent
2. Able to provide archival/fresh tumor tissues for biomarker analysis to assess PD-L1 expression and other biomarkers.
3. No known Epidermal Growth Factor Receptor (EGFR) or B-Raf proto-oncogene (BRAF) sensitizing mutation, or anaplastic lymphoma kinase (ALK) rearrangement or ROS proto oncogene 1 (ROS1) rearrangement
4. Radiographic progression per Response Evaluation Criteria in Solid Tumours (RECIST) v1.1 on or after anti-PD-(L)1 containing therapy for locally advanced and unresectable or metastatic NSCLC.
5. No prior anticancer therapy having the same mechanism of action as sitravatinib (eg, tyrosine kinase inhibitor with a similar target profile or vascular endothelial growth factor (VEGF)- or VEGFR inhibitor)
6. At least 1 measurable lesion as defined based on RECIST v1.1 by investigator

Key Exclusion Criteria:

1. Has received docetaxel as monotherapy or in combination with other therapies.
2. Squamous NSCLC with central cavitation, or NSCLC with hemoptysis (> 50 mL/day)
3. Participants with tumor shown by imaging to be located around important vascular structures or if the investigator determines that the tumor is likely to invade important blood vessels and may cause fatal bleeding.
4. Active leptomeningeal disease for metastatic NSCLC, or uncontrolled or untreated brain metastasis.
5. Active autoimmune diseases or history of autoimmune diseases that may relapse.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 377 (Actual)
Dates: Start 2021-07-27 (Actual); Primary Completion 2023-12-20 (Actual); Study Completion 2023-12-20 (Actual)

CONTACTS AND LOCATIONS:
Locations (61):
- Australia (9):
  - Blacktown Cancer and Haematology Centre, Blacktown, New South Wales
  - Campbelltown Hospital, Campbelltown, New South Wales
  - The Tweed Valley Hospital, Cudgen, New South Wales
  - St George Hospital, Kogarah, New South Wales
  - Pindara Private Hospital, Benowa, Queensland
  - Cancer Research South Australia, Adelaide, South Australia
  - Monash Health, Clayton, Victoria
  - St Vincents Hospital Melbourne, Fitzroy, Victoria
  - Sunshine Hospital, St Albans, Victoria
- China (52):
  - Anhui Provincial Cancer Hospital Aka West Branch of Anhui Province Hospital, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Peking Union Medical College Hospital, Beijing, Beijing Municipality
  - Xinqiao Hospital Affiliated to the Army Medical University, Chongqing, Chongqing Municipality
  - Daping Hospital, Third Military Medical University, Chongqing, Chongqing Municipality
  - Fujian Provincial Hospital, Fuzhou, Fujian
  - Fujian Cancer Hospital, Fuzhou, Fujian
  - The First Affiliated Hospital of Xiamen University, Xiamen, Fujian
  - The First Hospital of Lanzhou University, Lanzhou, Gansu
  - Cancer Center of Guangzhou Medical University, Guangzhou, Guangdong
  - Guangdong Provincial Peoples Hospital, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Cancer Hospital of Shantou University Medical College, Shantou, Guangdong
  - Cancer Hospital Chinse Academy of Medical Sciences, Shenzhen Center, Shenzhen, Guangdong
  - The Peoples Hospital of Guangxi Zhuang Autonomous Region, Nanning, Guangxi
  - The Tumor Hospital Affiliated to Guangxi Medical University, Nanning, Guangxi
  - Harbin Medical University Cancer Hospital, Harbin, Heilongjiang
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital of Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital of Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Hubei Cancer Hospital, Wuhan, Hubei
  - The Second Xiangya Hospital of Central South University, Changsha, Hunan
  - The First Peoples Hospital of Chenzhou, Chenzhou, Hunan
  - The Second Hospital, University of South China, Hengyang, Hunan
  - Changzhou No Peoples Hospital, the Affiliated Hospital of Nanjing Medical University Branch Cheng, Changzhou, Jiangsu
  - Nanjing First Hospital, Nanjing, Jiangsu
  - Zhongda Hospital Southeast University, Nanjing, Jiangsu
  - The Second Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - The Affiliated Hospital of Xuzhou Medical University, Xuzhou, Jiangsu
  - The First Affiliated Hospital of Nanchang University Branch Donghu, Nanchang, Jiangxi
  - The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi
  - The First Hospital of Jilin University, Changchun, Jilin
  - First Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - Liaoning Cancer Hospital and Institute, Shenyang, Liaoning
  - General Hospital of Ningxia Medical University, Yinchuan, Ningxia
  - Jinan Central Hospital, Jinan, Shandong
  - Shandong Cancer Hospital, Jinan, Shandong
  - The Affiliated Hospital of Qingdao University Branch Laoshan, Qingdao, Shandong
  - Rui Jin Hospital Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Affiliated Zhongshan Hospital of Fudan University, Shanghai, Shanghai Municipality
  - Huashan Hospital Affiliated to Fudan University, Shanghai, Shanghai Municipality
  - Sichuan Cancer Hospital and Institute, Chengdu, Sichuan
  - West China Hospital, Sichuan University, Chengdu, Sichuan
  - Tianjin Medical University General Hospital, Tianjin, Tianjin Municipality
  - Tianjin Medical University Cancer Institute and Hospital, Tianjin, Tianjin Municipality
  - Affiliated Cancer Hospital of Xinjiang Medical University, Ürümqi, Xinjiang
  - Yunnan Cancer Hospital, Kunming, Yunnan
  - Sir Run Run Shaw Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Zhejiang Cancer Hospital, Hangzhou, Zhejiang
  - Taizhou Hospital of Zhejiang, Taizhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Zhou Q, Zhao J, Gao B, et al. SAFFRON-301: A Phase 3 Study of Tislelizumab With Sitravatinib Versus Chemotherapy in Patients With Locally Advanced or Metastatic Non-Small Cell Lung Cancer Previously Treated With Platinum-Based Chemotherapy and an Anti-PD-1/PD-L1 Antibody. Poster presented at: ESMO Congress 2022; September, 2022; Paris, France.
- [Result] Zhou Q, Gao B, et al. SAFFRON-301: Sitravatinib PLUS Tislelizumab in Advanced/Metastatic NSCLC Progressing on/after Chemotherapy and Anti-PD-(L)1.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled across multiple study centers in China and Australia. The first participant was dosed on July 27th, 2021, and the last participant completed the study on December 20th, 2023. A decision to terminate the study was made on September 25th, 2023.
Pre-assignment Details: Patients were randomized in a 1:1 ratio to one of two treatment groups.
Groups:
- Tislelizumab + Sitravatinib: Participants received 200 mg of intravenous tislelizumab every 3 weeks, combined with 100 mg of oral sitravatinib daily.
- Docetaxel: Participants received 75 mg/m² of intravenous docetaxel every 3 weeks.
Period: Overall Study
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Started | 187 | 190
Treated | 186 | 177
Completed | 0 | 0
Not Completed | 187 | 190
Not completed — Withdrawal by Subject | 6 | 13
Not completed — Lost to Follow-up | 3 | 6
Not completed — Study Terminated by Sponsor | 86 | 89
Not completed — Death | 92 | 82

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) analysis set consists of all participants who were randomized to a treatment arm.
Groups:
- Total: Total of all reporting groups
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel | Total
Number analyzed (Participants) | 187 | 190 | 377
Age, Continuous [Mean (Standard Deviation); unit: Years] | 61.2 (8.43) | 61.3 (8.77) | 61.3 (8.60)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 34 | 39 | 73
  Male | 153 | 151 | 304
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 175 | 177 | 352
  White | 12 | 13 | 25
Region of Enrollment [Number; unit: participants]
  China | 174 | 175 | 349
  Australia | 13 | 15 | 28
Histology [Count of Participants; unit: Participants]
  Squamous | 96 | 97 | 193
  Non-squamous | 91 | 93 | 184
PD-L1 Expression Status [Count of Participants; unit: Participants] — Participants whose tissues were unevaluable for PD-L1 expression were included in the < 1% tumor cells group during randomization stratification.
  Participants
    >= 1% Tumor Cells | 71 | 71 | 142
    < 1% Tumor Cells | 116 | 119 | 235

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: Defined as the time from randomization until the date of death due to any cause. Kaplan-Meier methodology was used to estimate the median OS.
Time Frame: Until the study completion data cut-off date of December 20, 2023, or the last available date confirming participants were alive (a median follow-up of approximately 8 months).
Population: The Intent-to-Treat (ITT) analysis set consists of all participants who were randomized to a treatment arm.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 187 | 190
Months | 11.5 [9.4 to 14.6] | 11.4 [9.9 to 15.0]
Statistical Analysis 1: Comparison: Tislelizumab + Sitravatinib vs Docetaxel; Test type: Other; Hazard Ratio (HR) = 1.02, 95% CI 2-sided [0.75 to 1.39] — Hazard ratio and 95% confidence intervals (CIs) were estimated using a Cox regression model stratified by histological subtype (nonsquamous vs squamous), race (Asian vs Non-Asian) and PD-L1 expression (<1% Tumor Cells (TC) vs >=1% TC)

2. Primary Outcome: Progression Free Survival (PFS) as Assessed by the Independent Review Committee (IRC)
Description: Defined as the time from randomization until first documentation of disease progression as assessed by the IRC based on Response Evaluation Criteria in Solid Tumors (RECIST) v1.1, or death from any cause, whichever occured first. Kaplan-Meier methodology was used to estimate the median PFS.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 187 | 190
Months | 4.4 [4.0 to 5.7] | 2.9 [2.6 to 4.2]
Statistical Analysis 1: Comparison: Tislelizumab + Sitravatinib vs Docetaxel; Test type: Other; Hazard Ratio (HR) = 0.82, 95% CI 2-sided [0.62 to 1.07] — Hazard ratio and 95% CIs were estimated using a Cox regression model stratified by histological subtype (nonsquamous vs squamous), race (Asian vs Non-Asian) and PD-L1 expression (<1% TC vs >=1% TC)

3. Secondary Outcome: Progression Free Survival (PFS) as Assessed by the Investigator
Description: Defined as the time from randomization until first documentation of disease progression as determined by the investigator based on RECIST v1.1, or death from any cause, whichever occured first. Kaplan-Meier methodology was used to estimate the median PFS.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 187 | 190
Months | 4.4 [4.0 to 5.6] | 2.9 [2.6 to 4.1]
Statistical Analysis 1: Comparison: Tislelizumab + Sitravatinib vs Docetaxel; Test type: Other; Hazard Ratio (HR) = 0.64, 95% CI 2-sided [0.50 to 0.83] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Overall Response Rate (ORR)
Description: Defined as the percentage of participants with a confirmed complete response (CR) or partial response (PR) as assessed by the IRC per RECIST v1.1.
Time Frame: as for outcome 1
Population: ITT Analysis Set
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 187 | 190
percentage of participants | 12.3 [8.0 to 17.9] | 12.6 [8.3 to 18.2]

5. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the first occurrence of a documented objective response to the time of the first occurrence of disease progression, as determined by the IRC based on RECIST v1.1, or death from any cause, whichever occurs first.
Time Frame: as for outcome 1
Population: ITT Analysis Set. Only participants with best overall response of complete response or partial response confirmed per RECIST v1.1 were included in the analysis, and percentages were based on the number of responders.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 23 | 24
months | 6.0 [3.2 to 8.5] | NA [5.4 to NA] — Not estimable due to insufficient number of participants with events

6. Secondary Outcome: Disease Control Rate (DCR)
Description: Defined as the percentage of participants whose best overall response (BOR) is complete response, partial response, or stable disease per RECIST v1.1.
Time Frame: as for outcome 1
Population: ITT Analysis Set.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 187 | 190
percentage of participants | 69.5 [62.4 to 76.0] | 53.7 [46.3 to 60.9]

7. Secondary Outcome: Change From Baseline in European Organization for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30) Global Health Status (GHS) and Physical Functioning Scores
Description: The EORTC QLQ-30 contains 30 questions that incorporate 5 functional scales (physical functioning, role functioning, emotional functioning, cognitive functioning, and social functioning), 1 global health status scale, 3 symptom scales (fatigue, nausea and vomiting, and pain), and 6 single items (dyspnea, insomnia, appetite loss, constipation, diarrhea, and financial difficulties). The participant answers questions about their health during the past week. There are 28 questions answered on a 4-point scale where 1 = Not at all (best) and 4 = Very Much (worst) and 2 global health quality of life (QOL) questions answered on a 7-point scale where 1 = Very poor and 7 = Excellent. Raw scores are transformed into a 0 to 100 scale via linear transformation. Higher scores in GHS and functional scales indicate better quality of life.
Time Frame: Baseline and Cycle 5 Day 1 (Week 12) and Cycle 7 Day 1 (Week 18)
Population: Participants in the ITT Analysis Set with available at Baseline and each postbaseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 105 | 69
score on a scale
  Global Health Status at Cycle 5 | -5.5 (16.05) | -3.0 (18.69)
  Global Health Status at Cycle 7: number analyzed (Participants) | 84 | 52
  Global Health Status at Cycle 7 | -6.1 (15.86) | -3.4 (17.25)
  Physical Functioning at Cycle 5 | -4.1 (12.76) | -5.1 (15.89)
  Physical Functioning at Cycle 7: number analyzed (Participants) | 84 | 52
  Physical Functioning at Cycle 7 | -2.8 (12.30) | -3.1 (16.98)

8. Secondary Outcome: Change From Baseline in EORTC Quality of Life Questionnaire-Lung Cancer 13 (QLQ-LC13) Coughing, Dyspnoea, and Chest Pain Scales
Description: The EORTC QLQ-LC13 is the lung cancer module of the QLQ-C30 and measures lung cancer-specific disease and treatment symptoms. It includes 13 questions about specific symptoms in which participants respond based on a 4-point scale, where 1 is "not at all" and 4 is "very much". Raw scores are transformed into a 0 to 100 scale via linear transformation. Lower scores indicate an improvement in symptoms.
Time Frame: Baseline and Cycle 5 Day 1 (Week 12) and Cycle 7 Day 1 (Week 18)
Population: Participants in the ITT Analysis Set with available data at Baseline and each postbaseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 105 | 69
score on a scale
  Coughing at Cycle 5 | 1.6 (30.09) | -2.4 (27.61)
  Coughing at Cycle 7: number analyzed (Participants) | 84 | 52
  Coughing at Cycle 7 | -5.2 (25.08) | -1.3 (29.49)
  Dyspnoea at Cycle 5 | 2.6 (19.09) | 4.5 (16.76)
  Dyspnoea at Cycle 7: number analyzed (Participants) | 84 | 52
  Dyspnoea at Cycle 7 | -0.9 (14.66) | 2.1 (14.43)
  Chest Pain at Cycle 5 | -0.6 (24.45) | -0.5 (20.21)
  Chest Pain at Cycle 7: number analyzed (Participants) | 84 | 52
  Chest Pain at Cycle 7 | -2.4 (22.43) | -1.3 (16.12)

9. Secondary Outcome: Change From Baseline in European Quality of Life-5 Dimensions (EQ-5D-5L) Visual Analogue Scale (VAS)
Description: The EQ-5D-5L comprises a descriptive module that includes five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression and a Visual Analogue Scale. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The VAS records a participant's self-rated health on a vertical scale from 0 to 100, where 0 is 'the worst health you can imagine and 100 is 'the best health you can imagine'. A higher score indicates better health outcomes.
Time Frame: Baseline and Cycle 5 Day 1 (Week 12) and Cycle 7 Day 1 (Week 18)
Population: Participants in the ITT Analysis Set with available at Baseline and each postbaseline visit
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 105 | 69
score on a scale
  Cycle 5 | -6.1 (14.27) | -3.5 (13.76)
  Cycle 7: number analyzed (Participants) | 83 | 52
  Cycle 7 | -5.9 (12.31) | -3.2 (12.60)

10. Secondary Outcome: Number of Participants With Adverse Events
Description: Number of participants with treatment-emergent adverse events (TEAEs) and serious adverse events (SAEs), according to National Cancer Institute-Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Time Frame: From the first dose through 30 days after the final dose or until new anticancer therapy, whichever came first, (a median treatment duration of approximately 4 months in Arm 1 and 2 months in Arm 2).
Population: The Safety analysis set includes all participants who were randomized and received any dose of any study drug
Measure: Count of Participants; unit: Participants
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
Number analyzed (Participants) | 186 | 177
Participants
  TEAEs | 183 | 162
  SAEs | 83 | 66

ADVERSE EVENTS:
Time Frame: All-cause mortality is reported from randomization until the study completion data cut-off date of December 20, 2023, or the last available date confirming participants were alive ( a median follow-up of approximately 8 months). Adverse events are reported from the first dose through 30 days after the final dose or until new anticancer therapy, whichever came first, (a median treatment duration of approximately 4 months in Arm 1 and 2 months in Arm 2).
Description: All-cause mortality is reported for all randomized participants. Serious and other adverse events include all randomized participants who received ≥ 1 dose of any study treatment.
Arm/Group | Tislelizumab + Sitravatinib | Docetaxel
All-Cause Mortality (participants affected / at risk) | 92/187 | 82/190
Serious Adverse Events (participants affected / at risk) | 83/186 | 66/177
Other Adverse Events (participants affected / at risk) | 181/186 | 150/177
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Sitravatinib (N=186) | Docetaxel (N=177)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 7 (7)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 2 (2)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 8 (9)
Splenic infarction (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 1 (1) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Adrenal insufficiency (Endocrine disorders) | 2 (2) | 0 (0)
Immune-mediated hypophysitis (Endocrine disorders) | 1 (1) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0)
Ascites (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 2 (2)
Dysphagia (Gastrointestinal disorders) | 2 (2) | 1 (1)
Gastrointestinal perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1 (1) | 0 (0)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 2 (2) | 0 (0)
Oesophageal fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oesophageal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pancreatitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1)
Chest discomfort (General disorders) | 1 (1) | 1 (1)
Death (General disorders) | 6 (6) | 1 (1)
Fatigue (General disorders) | 3 (3) | 0 (0)
General physical health deterioration (General disorders) | 4 (4) | 2 (2)
Malaise (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Pyrexia (General disorders) | 1 (1) | 2 (2)
Drug-induced liver injury (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 3 (3) | 0 (0)
Immune-mediated hepatitis (Hepatobiliary disorders) | 4 (4) | 0 (0)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Biliary tract infection (Infections and infestations) | 1 (2) | 0 (0)
COVID-19 (Infections and infestations) | 2 (4) | 2 (2)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Febrile infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 2 (2) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1)
Infection (Infections and infestations) | 0 (0) | 1 (1)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 16 (16) | 17 (19)
Scrotal infection (Infections and infestations) | 1 (1) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 1 (1)
Radiation pneumonitis (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Alanine aminotransferase increased (Investigations) | 3 (3) | 2 (2)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0)
Electrocardiogram QT prolonged (Investigations) | 0 (0) | 1 (1)
Neutrophil count decreased (Investigations) | 0 (0) | 8 (8)
Platelet count decreased (Investigations) | 2 (2) | 1 (1)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 8 (8)
Decreased appetite (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypercalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (2) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 0 (0)
Hypoproteinaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Gouty arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Immune-mediated myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2)
Lymphangiosis carcinomatosa (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 0 (0)
Pericardial effusion malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Immune-mediated nephritis (Renal and urinary disorders) | 1 (1) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 1 (1)
Bronchopleural fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 6 (6)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 3 (3)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1)
Pulmonary infarction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 2 (2) | 0 (0)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Aortic dissection (Vascular disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2)
Shock (Vascular disorders) | 0 (0) | 1 (1)
Varicose vein (Vascular disorders) | 1 (1) | 0 (0)
Venous thrombosis limb (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tislelizumab + Sitravatinib (N=186) | Docetaxel (N=177)
Anaemia (Blood and lymphatic system disorders) | 61 (85) | 84 (163)
Leukopenia (Blood and lymphatic system disorders) | 0 (0) | 9 (18)
Neutropenia (Blood and lymphatic system disorders) | 2 (2) | 11 (18)
Thrombocytopenia (Blood and lymphatic system disorders) | 8 (11) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 8 (12) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 7 (10) | 7 (11)
Hypothyroidism (Endocrine disorders) | 46 (54) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 6 (7) | 3 (3)
Abdominal pain (Gastrointestinal disorders) | 14 (24) | 8 (14)
Abdominal pain upper (Gastrointestinal disorders) | 18 (23) | 3 (3)
Constipation (Gastrointestinal disorders) | 30 (33) | 26 (43)
Diarrhoea (Gastrointestinal disorders) | 82 (191) | 24 (37)
Dry mouth (Gastrointestinal disorders) | 6 (7) | 1 (1)
Mouth ulceration (Gastrointestinal disorders) | 6 (7) | 7 (8)
Nausea (Gastrointestinal disorders) | 29 (39) | 25 (40)
Stomatitis (Gastrointestinal disorders) | 12 (13) | 5 (6)
Vomiting (Gastrointestinal disorders) | 31 (45) | 19 (27)
Asthenia (General disorders) | 15 (16) | 15 (16)
Chest pain (General disorders) | 8 (9) | 1 (1)
Fatigue (General disorders) | 17 (18) | 17 (19)
Malaise (General disorders) | 5 (5) | 9 (12)
Non-cardiac chest pain (General disorders) | 3 (3) | 6 (6)
Oedema peripheral (General disorders) | 9 (10) | 6 (6)
Pain (General disorders) | 3 (3) | 6 (8)
Pyrexia (General disorders) | 18 (23) | 10 (19)
COVID-19 (Infections and infestations) | 10 (15) | 8 (17)
Pneumonia (Infections and infestations) | 10 (11) | 8 (8)
Upper respiratory tract infection (Infections and infestations) | 9 (11) | 6 (7)
Urinary tract infection (Infections and infestations) | 7 (9) | 2 (2)
Alanine aminotransferase increased (Investigations) | 96 (168) | 15 (15)
Alpha hydroxybutyrate dehydrogenase increased (Investigations) | 14 (21) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 111 (195) | 17 (21)
Bilirubin conjugated increased (Investigations) | 6 (8) | 5 (6)
Blood alkaline phosphatase increased (Investigations) | 26 (37) | 10 (15)
Blood bilirubin increased (Investigations) | 12 (18) | 6 (12)
Blood creatine phosphokinase MB increased (Investigations) | 74 (107) | 3 (3)
Blood creatine phosphokinase increased (Investigations) | 24 (32) | 6 (7)
Blood creatinine increased (Investigations) | 20 (29) | 8 (8)
Blood lactate dehydrogenase increased (Investigations) | 41 (74) | 8 (9)
Blood pressure increased (Investigations) | 7 (11) | 2 (3)
Blood thyroid stimulating hormone increased (Investigations) | 20 (20) | 1 (1)
Blood urea increased (Investigations) | 6 (15) | 2 (3)
Blood uric acid increased (Investigations) | 6 (16) | 1 (1)
C-reactive protein increased (Investigations) | 5 (6) | 6 (6)
Electrocardiogram QT prolonged (Investigations) | 7 (10) | 1 (1)
Gamma-glutamyltransferase increased (Investigations) | 27 (41) | 13 (16)
Lymphocyte count decreased (Investigations) | 9 (13) | 19 (54)
Neutrophil count decreased (Investigations) | 10 (12) | 54 (162)
Neutrophil count increased (Investigations) | 6 (12) | 4 (5)
Platelet count decreased (Investigations) | 36 (58) | 22 (47)
Protein urine present (Investigations) | 14 (19) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 23 (26) | 10 (11)
Weight decreased (Investigations) | 54 (65) | 15 (17)
White blood cell count decreased (Investigations) | 11 (17) | 62 (201)
White blood cells urine positive (Investigations) | 6 (6) | 2 (4)
Decreased appetite (Metabolism and nutrition disorders) | 53 (62) | 29 (33)
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 (17) | 5 (6)
Hyperglycaemia (Metabolism and nutrition disorders) | 15 (22) | 18 (24)
Hyperlipidaemia (Metabolism and nutrition disorders) | 7 (10) | 2 (2)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 19 (35) | 5 (8)
Hyperuricaemia (Metabolism and nutrition disorders) | 19 (39) | 8 (14)
Hypoalbuminaemia (Metabolism and nutrition disorders) | 57 (85) | 41 (60)
Hypocalcaemia (Metabolism and nutrition disorders) | 27 (40) | 13 (31)
Hypochloraemia (Metabolism and nutrition disorders) | 9 (13) | 3 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 35 (53) | 15 (28)
Hypomagnesaemia (Metabolism and nutrition disorders) | 7 (14) | 3 (5)
Hyponatraemia (Metabolism and nutrition disorders) | 43 (72) | 18 (22)
Hypophosphataemia (Metabolism and nutrition disorders) | 9 (11) | 3 (9)
Hypoproteinaemia (Metabolism and nutrition disorders) | 6 (6) | 3 (3)
Arthralgia (Musculoskeletal and connective tissue disorders) | 6 (8) | 10 (10)
Back pain (Musculoskeletal and connective tissue disorders) | 12 (16) | 7 (10)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 9 (9) | 11 (11)
Headache (Nervous system disorders) | 9 (10) | 8 (8)
Hypoaesthesia (Nervous system disorders) | 4 (4) | 7 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 1 (1) | 9 (10)
Insomnia (Psychiatric disorders) | 20 (25) | 14 (15)
Haematuria (Renal and urinary disorders) | 14 (18) | 4 (14)
Proteinuria (Renal and urinary disorders) | 34 (55) | 13 (18)
Cough (Respiratory, thoracic and mediastinal disorders) | 26 (29) | 28 (31)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 25 (26) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13 (13) | 12 (12)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 25 (33) | 18 (20)
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 10 (12) | 4 (4)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 9 (9)
Alopecia (Skin and subcutaneous tissue disorders) | 5 (5) | 59 (60)
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 67 (76) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 8 (8) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 32 (41) | 10 (11)
Hypertension (Vascular disorders) | 56 (65) | 6 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
BeiGene has 18 months from the end of the study at all sites to publish overall study results. After the 1st multi-site publication or the expiration of publication period, Investigators are free to publish/present the results of the study. Investigators must submit all draft publications/presentations to us for review 60 days prior to the planned publication/presentation date. BeiGene may request deletion of its confidential information & may request a further delay to protect its IP rights.

DOCUMENTS (2):
  • Study Protocol (2022-08-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04921358/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-09): https://cdn.clinicaltrials.gov/large-docs/58/NCT04921358/SAP_001.pdf